CLINICAL TRIAL: NCT04197076
Title: An Open, Observational Clinical Study, 2-3 Cycles Treatment as Neoadjuvant Therapy for NSCLC With Stage IIB-IIIB
Brief Title: Neoadjuvant Therapy in Resectable Non-Small Cell Lung Cancer Stages IIB-IIIB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Lu Shun, Director of Oncology, Shanghai Chest Hospital
Other Study IDs: Neoadjuvant study of NSCLC
Record Dates: First submitted 2019-04-27; First posted 2019-12-12 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subject's tumor sample obtained within 3 months before enrollment is suitable to be used for gene testing（EGFR/ALK/ROS1）and PD-L1 testing with Immunohistochemistry (IHC)。
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neoadjuvant immunotherapy: pd-1 or pd-l1 inhabitors
  Interventions: Drug: anti-PD-1 or anti-PD-L1
- Neoadjuvant targeted therapy: TKIs
  Interventions: Drug: EGFR-TKI, ALK inhibitor, ROS1 inhibitor
- Neoadjuvant chemotherapy: chemotherapy
  Interventions: Drug: investigator decided

INTERVENTIONS:
Drug: anti-PD-1 or anti-PD-L1 — immunotherapy anti-PD-1 or anti-PD-L1
  Other Names: Neoadjuvant immunotherapy
  Groups: Neoadjuvant immunotherapy
Drug: EGFR-TKI, ALK inhibitor, ROS1 inhibitor — targeted therapy EGFR-TKI, ALK inhibitor, ROS1 inhibitor
  Other Names: Neoadjuvant targeted therapy
  Groups: Neoadjuvant targeted therapy
Drug: investigator decided — chemotherapy
  Other Names: Neoadjuvant chemotherapy
  Groups: Neoadjuvant chemotherapy

SUMMARY:
This study aims to investigate the efficacy and safety of targeted therapy and chemotherapy±immunotherapy as neoadjuvant therapy in stage IIB-IIIB NSCLC patients.（observational study）

DETAILED DESCRIPTION:
This is an open, observational clinical study, 2-3 cycles treatment will be planned as neo-adjuvant therapy for NSCLC participants in stage IIB-IIIB.

Study design:

Newly diagnosed Resectable IIB-IIIB NSCLC EGFR/ALK/ROS1 TEST PD-L1 TEST Collect puncture biopsy tissue/ Blood sample in screening period Chest enhanced CT Conditions allowed， whole body PETCT Exam; Group A：Targeted therapy Tumors with Driver genes （EGFR/ALK/ROS1 Positive） 2 cycles（42 days; Group B：Immunotherapy Enroll Patients from 816 Research treated with Neoadjuvant immunotherapy Or, treated with immunotherapy in practice（with approval） Group C：Routine Chemotherapy Driver genes（EGFR/ALK/ROS1 Negative） and PD-L1 Test negative or unknown; Operation （within 6 Ws postoperation） Standard treatment， Allow adjuvant chemotherapy±radio therapy Collect resected tissue sample(Tumor T and Node N) /Blood sample; comparisons before and after treatment: Imaging：CT、PET-CT Sample：Tumor tissue、blood

Objective and End point:

1. Main objective and end point：DFS，pCR rate
2. Second objective and end point：OS
3. Exploratory objective and end point：cRR rate、relevant AE、Change of Scoring Scale、exploration for relevant biological indicators

ELIGIBILITY:
Inclusion Criteria:

1. Primary non-small cell lung cancer confirmed by cytology or histology
2. According to the TNM stage (8th Edition) of IASLC lung cancer, it is determined to be IIB-IIIB stage non-small cell lung cancer, which is considered to be resectable;
3. There must be at least one evaluable focus judged according to recist1.1 standard (the longest diameter on spiral CT is at least 10 mm, and the longest diameter on general CT is at least 20 mm)
4. ECOG PS 0 or 1
5. There are tumor samples available for gene detection (EGFR / ALK / ros1) and PD-L1 immunohistochemistry (IHC) in the subjects, and the tumor samples should be obtained within 3 months before enrollment.
6. If all suspected mediastinal lymph nodes (including those with pathological enlargement or FDG concentration on PET / CT) can be examined by EBUS, thoracoscopy or mediastinoscopy, further sampling is required for pathological confirmation.
7. Male or female, ≥ 18 years old
8. Adequate blood function: absolute neutrophil count (ANC) ≥ 2 × 109 / L, platelet count ≥ 100 × 109 / L and hemoglobin 110 ≥ 9 g / dl
9. Adequate liver function: total bilirubin ≤ upper limit of normal value (ULN); AST and alt ≤ upper limit of normal value (ULN); alkaline phosphatase ≤ upper limit of normal value (ULN)
10. Adequate renal function: serum creatinine ≤ upper limit of normal value (ULN) or calculated creatinine clearance ≥ 60ml / min
11. No anti-tumor drug treatment in the past
12. For patients who have had previous surgery, it is required that more than 4 weeks have passed since the start of study treatment, and the patients have recovered
13. Women with a full uterus must have negative pregnancy test results within 28 days before entering the study (unless it is 24 months after amenorrhea). If the pregnancy test is more than 7 days from the first administration, a urine pregnancy test is required for verification (within 7 days before the first administration)
14. Sign the informed consent form (the informed consent form needs to be approved by the independent ethics committee, and the informed consent of the patient should be obtained before starting any substantive trial procedure)

Exclusion Criteria:

1. Have other malignant tumors in the last 5 years
2. AST and / or ALT > 2.5 times of the upper limit of normal value (ULN), with alkaline phosphatase > 5 times of the upper limit of normal value (ULN)
3. Previously received radiotherapy
4. Previously used chemotherapy drugs, targeted and immunotherapy drugs (except bisphosphonates)
5. There are any uncontrolled systemic diseases, including active infection, uncontrolled hypertension, diabetes, unstable angina, congestive heart failure, myocardial infarction (within 1 year before treatment), serious arrhythmia requiring drug treatment, liver, kidney and metabolic diseases
6. Women in pregnancy or lactation
7. The patient (male or female) has the possibility of childbearing but is unwilling or does not take effective contraceptive measures
8. Receive the experimental treatment of other clinical studies at the same time (in the treatment period of clinical studies)
9. Known to be allergic to possible chemotherapy drugs
10. There is evidence of other diseases, neurological or metabolic dysfunction, abnormal physical examination or laboratory examination, and it is suspected that there may be a high risk of contraindications to the study drug or complications related to treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC participants in stage IIB-IIIB(American Joint Committee on Cancer 8th edition criteria)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
DFS: disease free survival | 36 months
  The time length from randomization(mainly from the receipt of pathology and genetic diagnosis reports)to any of the following events: disease progression, disease recurrence or death from any cause. Disease progression or relapse will be assessed according to RECIST 1.1
pCR: pathologic complete response | 36 months
  the proportion of patients achieved pathologic complete response（lung and lymph node without tumor residual assessed by pathology review)

SECONDARY OUTCOMES:
OS: Overall survival | 36 months
  The time length from the date of randomization (according to the received pathology and genetic diagnosis report) to the date of death.

OTHER OUTCOMES:
cRR rates | approximately 10 weeks After surgery
  The proportion of patients achieved complete or patial remission(Imageological) according to RECIST 1.1 prior to definitive surgery
Safty AEs | 36 months
  proportion of delayed or cancelled surgery or duration of surgery or length of hospitalization or surgical procedure, and incidence of AE/SAE associated with surgery, Adverse events will be graded according to NCI CTCAE
Qol Quality of Life | 36 months
  Quality of life asscesed by Quality of Life Questionnare-Core 30(EORTC QLQ-C30）of The European O-rganization for Reasearch and Treatment of Cancer containing 30 items in total. Among them, items 29 and 30 are divided into seven grades. According to the answer options 1 to 7 points. Other items are divided into four grades: none, one point, some to many. When scoring, they are directly rated 1 to 4 points. For functional and overal health domain, higher score means better life quality; for symptom domain ,higher score means worse life quality.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Study Chair — Shanghai Chest Hospital
Locations (1):
- Oncology Department, Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qi Y, Gu L, Shen J, Yao Y, Zhao Y, Lu S, Chen Z. An open, observational clinical study of neoadjuvant therapy in resectable stage III non-small cell lung cancer. Front Oncol. 2023 Aug 16;13:1194100. doi: 10.3389/fonc.2023.1194100. eCollection 2023. PMID 37655106
- [Derived] Gu L, Wang X, Sun Y, Xu Y, Niu X, Zhao R, Yao Y, Jian H, Han Y, Wei J, Chen Z, Lu S. An open, observational, three-arm clinical study of 2-3 cycles of treatment as neoadjuvant therapy in operable locally advanced non-small cell lung cancer: An interim analysis. Front Immunol. 2022 Aug 19;13:938269. doi: 10.3389/fimmu.2022.938269. eCollection 2022. PMID 36059450